CLINICAL TRIAL: NCT06151210
Title: A Multicenter, Randomized, Double-blind, Active-controlled, Parallel, Phase III Clinical Trial to Evaluate the Efficacy and Safety of DA-5219 in Patients With Acute or Chronic Gastritis
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety of DA-5219 in Patients With Acute or Chronic Gastritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DA5219_GAS_III
Record Dates: First submitted 2023-11-21; First posted 2023-11-30 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Gastritis Acute; Gastritis Chronic
MeSH Terms: interventions — DA 9601

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DA-5219 (Experimental): administered for 2weeks(DA-5219 + Stillen® Tab placebo)
  Interventions: Drug: DA-5219; Drug: Stillen® Tab Placebo
- Stillen® Tab (Active Comparator): administered for 2weeks(Stillen® Tab + DA-5219 placebo)
  Interventions: Drug: Stillen® Tab; Drug: DA-5219 Placebo

INTERVENTIONS:
Drug: DA-5219 — 1 tablet/day
  Arms: DA-5219
Drug: Stillen® Tab — 3 tablets/day
  Arms: Stillen® Tab
Drug: DA-5219 Placebo — 1 tablet/day
  Arms: Stillen® Tab
Drug: Stillen® Tab Placebo — 3 tablets/day
  Arms: DA-5219

SUMMARY:
This study is to evaluate the efficacy and safety of DA-5219 in patients with acute or chronic gastritis

ELIGIBILITY:
Main Inclusion Criteria:

* Men or women aged ≥ 19 years and ≤ 75 years
* Subjects who diagnosed with acute or chronic gastritis by upper gastrointestinal endoscopy within 7days prior to the randomization
* Subjects who have one or more erosions identified on upper gastrointestinal endoscopy within 7days prior to the randomization
* Subjects who voluntarily signed a consent form

Main Exclusion Criteria:

* Ineligible for upper gastrointestinal endoscopy
* Subjects with active or healing gastroduodenal ulcer, reflux esophagitis, Barrett's esophagus, or gastroesophageal varices identified on upper gastrointestinal endoscopy within 7days prior to the randomization
* Subjects with hypersensitivity to investigational drugs and similar drugs
* Pregnant or breastfeeding women

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 467 (Actual)
Dates: Start 2024-01-31 (Actual); Primary Completion 2025-07-10 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Improvement rate of gastric mucosal erosion | Change from baseline at 2 weeks

SECONDARY OUTCOMES:
Cure rate for gastric mucosal erosion | Change from baseline at 2 weeks
Cure rate for gastric mucosal edema | Change from baseline at 2 weeks
Improvement rate for gastric mucosal erythema | Change from baseline at 2 weeks
Improvement rate for gastric mucosal bleeding | Change from baseline at 2 weeks
Improvement rate for gastric subjective symptoms | Change from baseline at 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes